CLINICAL TRIAL: NCT00299520
Title: Phase 3, Randomized, Investigator-Blind, Multi-Center Study to Evaluate Efficacy and Safety of Intravenous Iclaprim Versus Linezolid in Complicated Skin and Skin Structure Infections.(ASSIST-1)
Brief Title: Phase 3 Safety and Efficacy Study of I.V. Iclaprim v Linezolid in cSSSI (ASSIST-1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arpida AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol No. ICLA-08-CSI1; ASSIST-1
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: Complicated Skin and Skin Structure Infection
Keywords: skin infection; complicated skin infection; skin structure infection
MeSH Terms: conditions — Cellulitis

INTERVENTIONS:
Drug: intravenous iclaprim or intravenous linezolid

SUMMARY:
This is a multi-center, investigator-blind, comparative Phase 3 study. Patients will receive either iclaprim or linezolid for 10 to 14 days. Patients will be evaluated daily for the first four days of study treatment and then every other day, for up to 14 days of the treatment period, at End of Therapy, the Test Of Cure visit (7 to 14 days post treatment), and a Late Follow-up (F/U) visit (7 to 14 days after the TOC visit).

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of this study is to compare the clinical cure rates of iclaprim and linezolid at the test of cure (TOC) visit (7 to 14 days after the end of treatment).

Secondary Objectives:

The secondary objectives of this study are to compare iclaprim with linezolid regarding:

* Clinical efficacy at the end of study medication treatment;
* Time to resolution of systemic and local signs and symptoms of complicated skin and skin structure infection (cSSSI);
* Clinical outcome in the microbiologically evaluable (ME) population;
* Bacteriologic outcome in the ME population;
* Bacteriologic eradication rates of Baseline (BL) pathogens;
* Clinical outcome in the modified intent-to-treat (MITT) population;
* Bacteriologic outcome in the MITT population;
* Baseline in vitro susceptibility of isolated pathogens in the ME population; and
* Safety and tolerability of iclaprim treatment.

ELIGIBILITY:
Inclusion Criteria -Diagnosis of an infection consistent with complicated skin and skin structure infection due to a gram positive pathogen.

Exclusion Criteria: - Known or suspected hypersensitivity to any study medication or other related anti-infective medication - Any known or suspected condition or concurrent treatment contraindicated by the prescribing information - Previous enrollment in this study - Treatment with any investigational drug within 30 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-06; Study Completion 2006-07

PRIMARY OUTCOMES:
Clinical cure rate (the ratio of number of clinically cured patients to the total number of patients in the population) at 7 to 14 days after the end of therapy

SECONDARY OUTCOMES:
Microbiological eradication rate at 7-14 days after end of therapy.
Safety evaluations conducted during the study

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - e-Study Site, National City, California
  - VA Medical Center, Boise, Idaho
  - Infectious Disease of Indiana, Indianapolis, Indiana
  - Judith Stone. M.D., Cumberland, Maryland
  - ID Clinical Research, Ltd., Toledo, Ohio

REFERENCES:
- See also: ARPIDA AG corporate website — http://www.arpida.ch